CLINICAL TRIAL: NCT01932710
Title: A Feasibility Study of White Blood Cell Transfusion for the Prevention of Infection in Acute Myelogenous Leukemia Patients Undergoing Front-Line or First Salvage Induction Therapy
Brief Title: A Feasibility Study of Prophylactic White Blood Cell Transfusions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012-1158; NCI-2013-02208 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Leukemia
Keywords: Leukemia; Acute myelogenous leukemia; AML; High-risk myelodysplastic leukemia; MDS; Infection risk; White Blood Cell transfusion; Prophylactic therapy
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Leukocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- White Blood Cell Transfusion (Experimental): Patient receives white blood cells by vein from a volunteer donor. Each transfusion will take anywhere from 1 hour to several hours, depending on how treatment is tolerated. Patient receives a transfusion every 3-4 days (at least 2 a week) for up to 6 weeks.
  Interventions: Procedure: White Blood Cell Transfusion

INTERVENTIONS:
Procedure: White Blood Cell Transfusion — Patient receives white blood cells by vein from a volunteer donor. Each transfusion will take anywhere from 1 hour to several hours, depending on how treatment tolerated. Transfusion received every 3-4 days (at least 2 a week) for up to 6 weeks.

SUMMARY:
Patients with leukemia often have low white blood cell counts after chemotherapy, which puts them at greater risk of infection. The standard of care for preventing infections is to give these patients antibiotic, antifungal, and antiviral drugs during the time that white blood cell counts are low. However, many patients still develop infections during chemotherapy. Radiated white blood cell transfusions are a standard treatment once a patient develops a severe infection.

The goal of this clinical research study is to learn if giving white blood cell transfusions that are not radiated early in chemotherapy might delay or prevent infections in patients with leukemia. Researchers also want to learn more about the type and severity of any infections that do occur.

DETAILED DESCRIPTION:
Study Procedures:

During each white blood cell transfusion, you will receive white blood cells from a volunteer donor through a needle in your vein. Each transfusion will take anywhere from 1 hour to several hours, depending on how you tolerate the treatment. You will receive a transfusion approximately every 3-4 days (2 a week) for up to 6 weeks.

Before each white blood cell transfusion, your vital signs (temperature, heart rate, breathing rate, and blood pressure) will be recorded according to standard evaluation of patients with fever to look for underlying infectious causes. During and for 1 hour after the transfusion, you will be monitored for side effects. You may be given a drug to help or reduce any side effects. Your doctor will tell you more about any drug that may be given for side effects.

If at any point you develop a fever while on study, blood (about 1 teaspoon) and urine will be collected to check for infection according to standard evaluation of patients with fever to look for underlying infectious causes. You may also have a chest x-ray. If it is abnormal or if you have symptoms (cough, shortness of breath, nasal congestion), you may need a computed tomography (CT) scan of the chest and/or sinuses. That will be done within 3 days of developing a fever. If the doctor thinks it is needed, you will than have another CT scan 2 weeks later and at any other point that the doctor thinks it are needed to check for infection.

Length of Study:

You will continue to have transfusions until the doctor thinks infection has been controlled or until your white blood cell counts stay at a certain level for at least 2 days in a row. If any point you are discharged from the hospital and your doctor wants you to continue receiving white blood cell transfusions, you will be able to receive them as an outpatient.

You will be monitored for side effects and signs of infection for up to 6 weeks. You will be taken off study if you have intolerable side effects.

This is an investigational study. Radiated white blood cell transfusions are considered to be a standard procedure for the treatment of serious infections. It is investigational to give unirradiated white blood cell transfusions as a way of preventing infections.

Up to 50 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. All acute myelogenous leukemia and high-risk myelodysplastic leukemia patients who are admitted to the leukemia service and those who are referred from other services (i.e. pediatrics, medical oncology, etc.) will be eligible for the study.
2. Patients will be undergoing initial therapy for their disease or undergoing first salvage treatment, i.e. patients who fail therapy, or respond and relapse after initial therapy.
3. Patients will be free of signs and symptoms of infection at the time of entering the study and, most importantly, will be encouraged to have sufficient donors to administer prophylactic white cell transfusion twice a week for six weeks in order to assess their effectiveness.

Exclusion Criteria:

1. Patients with baseline (at start leukemia treatment) infection, defined as patients with a) fever and known positive cultures at the time of registration; or b) chest or sinus computed tomography with findings suggestive of pneumonia or sinusitis; or c) one positive galactomannan test >/= 1 or two positive galactomannan text >/= 0.5 to 1.
2. Patients with Zubrod performance status >/= 3.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Utilizing White Cell Transfusion as a Prophylactic Therapy | 6 weeks
  Study considered feasible if within one year, 20 patients enrolled with sufficient donors to donate white blood cells, two transfusion per week for six weeks (on average a total of 12 white blood transfusions per patient) to participate in the prophylactic therapy.

SECONDARY OUTCOMES:
Infection Rate | 6 weeks
  For the secondary analysis, the infection rate with its 95% CI will be estimated for patients with and without sufficient donors, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org